CLINICAL TRIAL: NCT03866980
Title: A Phase III, Randomized, Double-blinded, Multicenter Study of AK105 Combined With Carboplatin and Pemetrexed vs Placebo Combined With Carboplatin and Pemetrexed as First-line Therapy in Patients With Metastatic Nonsquamous Non-small Cell Lung Cancer
Brief Title: A Study of Anti-PD-1 AK105 in Patients With Metastatic Nonsquamous Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: corporate strategy adjustment
Sponsor: Akeso (Industry)
Collaborators: Akeso Tiancheng, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK105-301
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer Non-small Cell Stage IV
Keywords: immunotherapy,immuno-oncology, non-small cell lung cancer; Anti-PD-1 antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AK105 plus Carboplatin and Pemetrexed (Experimental): Subjects receive AK105 200 mg intravenously (IV) plus pemetrexed 500 mg/m^2 IV and carboplatin area under the curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK105 200 mg IV plus pemetrexed 500 mg/m^2 IV Q3W until progression.
  Interventions: Biological: AK105; Drug: carboplatin; Drug: pemetrexed
- Placebo plus Carboplatin and Pemetrexed (Placebo Comparator): Subjects receive placebo intravenously (IV) plus pemetrexed 500 mg/m^2 IV and carboplatin area under the curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK105 200 mg IV plus pemetrexed 500 mg/m^2 IV Q3W until progression.
  Interventions: Drug: carboplatin; Drug: pemetrexed; Drug: placebo
- AK105 plus anlotinib (Experimental): Subjects receive AK105 200 mg intravenously (IV) plus Anlotinib 12mg/d PO D1-14, Q3W until progression.
  Interventions: Biological: AK105; Drug: Anlotinib

INTERVENTIONS:
Biological: AK105 — IV infusion
  Arms: AK105 plus Carboplatin and Pemetrexed; AK105 plus anlotinib
Drug: carboplatin — IV infusion
  Arms: AK105 plus Carboplatin and Pemetrexed; Placebo plus Carboplatin and Pemetrexed
Drug: pemetrexed — IV infusion
  Arms: AK105 plus Carboplatin and Pemetrexed; Placebo plus Carboplatin and Pemetrexed
Drug: placebo — IV infusion
  Arms: Placebo plus Carboplatin and Pemetrexed
Drug: Anlotinib — PO
  Arms: AK105 plus anlotinib

SUMMARY:
This is a phase III , randomized, double-blinded, multicenter clinical study to compare efficacy and safety of AK105 (Anti-PD1 antibody) combined with Carboplatin and Pemetrexed vs Placebo combined with Carboplatin and Pemetrexed as first-line therapy in patients with EGFR and ALK wild type metastatic nonsquamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Age over 18 years old (inclusive) and not more than 75 years old (inclusive), when signing the ICF.
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Expected life expectance ≥ 3 months.
* Histologically or cytologically confirmed diagnosis of stage IV nonsquamous NSCLC.
* No prior systemic chemotherapy for advanced or metastatic NSCLC. Subjects who have received prior adjuvant chemotherapy or neoadjuvant chemotherapy with curative intent, or definitive chemoradiotherapy for advanced disease, will be eligible provided that progression has occurred >6 months from last treatment.
* At least one measurable tumor lesion per RECIST 1.1 criteria. A lesion previously irradiated will not be considered a target lesion.
* Subjects must provide an available tumor tissue sample taken < 12 months prior to first dose of study treatment.
* Subjects must provide wild-type EGFR and ALK reported by tissue-based tests. For subjects without documented wild-type EGFR/ALK, archival or fresh tumor tissues are required for EGFR/ALK assessment prior to enrollment.
* Adequate organ function.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.

Exclusion Criteria:

* Subjects who are diagnosed as NSCLC that harbors an EGFR-sensitizing mutation or ALK gene translocation.
* Subjects with other histological types of NSCLC, including mixed squamous cell carcinoma and adenocarcinoma, and mixed carcinoma containing small cell lung carcinoma or neuroendocrine carcinoma.
* Received prior treatment with EGFR inhibitors or ALK inhibitors.
* Receipt of last radiotherapy or any anti-tumor treatment [chemotherapy, targeted therapy, immunotherapy, Chinese patent drugs with antitumor indications, or immunomodulators or tumor embolization] within 3 weeks prior to the first dose of study treatment.
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (e.g. CD40, CD137, GITR and OX40 etc).
* Other invasive malignancies within 5 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
* Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
* Active or previously documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea).
* Subjects who require systemic corticosteroids (a dose equivalent to >10 mg/day prednisone) or other immunosuppressive drugs within 14 days prior to the first dose of study drug.
* Major surgery (as defined by the investigator) within 28 days prior to the first dose of study drug.
* Subjects who received non-thoracic radiotherapy >30 Gy within 4 weeks prior to the first dose, or thoracic radiotherapy >30 Gy within 24 weeks prior to the first dose study drug.
* History of gastrointestinal perforation and/ or fistula within 6 months prior to the first dose of study drug.
* Known history of primary immunodeficiency virus infection.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Known history of interstitial lung disease.
* Known history of active tuberculosis (TB).
* An active infection requiring systemic therapy.
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Known history of testing positive for human immunodeficiency virus (HIV).
* Presence of meningeal metastasis, spinal cord compression, leptomeningeal disease or active brain metastasis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Clinically active hemoptysis, active diverticulitis, peritoneal abscess, or gastrointestinal obstruction.
* Clinically significant bleeding symptoms or significant bleeding tendency such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis within 1 month prior to the first dose of study treatment.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria, with the exception of alopecia.
* Receipt of live or attenuated vaccination within 30 days prior to the first dose of study treatment, or plan to receive live or attenuated vaccine during the study.
* Known history of server hypersensitivity to other monoclonal antibodies.
* Known severe allergic reactions to anlotinib,pemetrexed, carboplatin or platinum-containing component, or their preventive medications.
* Known allergic reactions to any ingredients of AK105.
* Pregnant or lactating women.
* Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in intent-to-treat (ITT) population, assessed by Independent Radiologist Review Committee(IRRC) in accordance with RECIST v1.1 | up to 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by IRRC or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
Overall survival (OS) in ITT population | Up to 2 years
  OS is the time from the date of randomization to death due to any cause.
PFS assessed by the investigator in accordance with RECIST v1.1 | Up to 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Objective response rate (ORR) | Up to 2 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1.
Duration of response (DoR) | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST v1.1.
Incidence and severity of treatment-emergent adverse events (TEAEs) | From the time of informed consent signed through 90 days after last dose of AK105
  An adverse event (AE) is any untoward medical occurrence or the deterioration of existing medical event in a clinical study subject administered an investigational drug, which does not necessarily have an unequivocal causal relationship with the investigational product.
Observed concentrations of AK105 | From first dose of AK105 through 90 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through 90 days after last dose of AK105
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Shunchang Jiao, MD, Study Chair — Chinese PLA General Hospital; Baohui Han, MD, Study Chair — Shanghai Chest Hospital
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Pang X, Zhong T, Qu T, Chen N, Ma S, He X, Xia D, Wang M, Xia M, Li B. Penpulimab, an Fc-Engineered IgG1 Anti-PD-1 Antibody, With Improved Efficacy and Low Incidence of Immune-Related Adverse Events. Front Immunol. 2022 Jun 27;13:924542. doi: 10.3389/fimmu.2022.924542. eCollection 2022. PMID 35833116